CLINICAL TRIAL: NCT01378260
Title: Comparative Effectiveness Research Study of Peripheral Arterial Disease (PAD)
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, David Flum, Professor, University of Washington
Other Study IDs: 40153; R01HS2002501
Record Dates: First submitted 2011-06-13; First posted 2011-06-22 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Arterial Disease; Claudication
Keywords: Peripheral Arterial Disease; Claudication; Comparative Effectiveness Research; PAD Study; PAD; atherosclerosis; Intermittent claudication; leg pain
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Surgical Bypass: use of synthetic or endogenous (vein) or composite graft to treat lesions in the superficial femoral, common femoral, or popliteal artery
- Endovascular Therapy: angioplasty and/or stent to treat lesions in the superficial femoral or popliteal artery
- Medical Management: Documentation of the following in the medical record:
  i. Walking/physical therapy to improve endurance was recommended; ii. For tobacco users, tobacco cessation was recommended; iii. Prescribing pentoxifylline (Trental) or cilostazol (pletal) iv. Ongoing care by physician for treatment of claudication

SUMMARY:
The specific aim of this study is to prospectively compare outcomes (functional, quality of life, risk-adjusted clinical event) of medical management, surgical or endovascular (angioplasty or stent placement) interventions for the treatment of claudication caused by peripheral arterial disease. This study will test two major hypotheses;

Hypothesis 1: At 12-months, surgical interventions are associated with greater improvements in function, claudication symptoms, and health-related quality of life (HRQoL) than endovascular procedures or medical management.

Hypothesis 2: At 12-months, surgical and endovascular interventions are associated with greater improvements in function, claudication symptoms, and HRQoL than medical management.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of claudication
2. Be undergoing one of three treatments for claudication:

   * Surgical bypass (use of synthetic or endogenous (vein) or composite graft to treat lesions in the superficial femoral, common femoral or popliteal artery)
   * Endovascular therapy (angioplasty and/or stent to treat lesions in the superficial femoral, common femoral or popliteal artery)
   * Medical management (i.e. smoking cessation, walking therapy, long-term monitoring by physician)

Exclusion Criteria:

1. those with documented acute ischemia, rest pain or ulceration
2. those with claudication determined to be of aortic or iliac origin
3. those with claudication that is not caused by atherosclerotic disease
4. those without access to a telephone or Internet and are unwilling to participate in surveys by mail at home (assess in patient screen)
5. those who otherwise refuse to participate (assessed in patient screen)
6. those who have a diagnosis of dementia confirmed in their medical record
7. those who are not English speaking
8. children and young adults up to and including age 20-years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients being seen by a physician with newly diagnosed or established claudication
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in score on the Walking Impairment Questionnaire (WIQ) from the baseline assessment to the 12-month assessment. | 12-Months Post-Index Date
  The primary outcome of the study, and the outcome on which the study is powered, is the change in score on the WIQ from the baseline assessment to the 12-month assessment. There are three subscales within the WIQ; summary scores will be calculated separately for each - the walk distance, walk speed, stair climb.

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, Principal Investigator — University of Washington
Locations (12):
- United States (12):
  - Lake Washington Vascular, Bellevue, Washington
  - PeaceHealth St. Joseph Medical Center, Bellingham, Washington
  - Providence Everett, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Good Samaritan Hospital, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Northwest Hospital and Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - St. Joseph Medical Center, Tacoma, Washington
  - Tacoma General Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center - Thoracic & Vascular Surgery, Vancouver, Washington